CLINICAL TRIAL: NCT03819907
Title: The Use of Virtual Reality for Lumbar Pain Management in an Outpatient Spine Clinic: An Exploratory Comparative Randomized Trial
Brief Title: The Use of Virtual Reality for Lumbar Pain Management in an Outpatient Spine Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, David Saul Binder, Director of Innovation, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P003042Final
Record Dates: First submitted 2019-01-17; First posted 2019-01-29 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 15 participants will be randomly assigned to the control group. They will receive no intervention other than the injection (which is not a part of the trial).
  Pre-injection they will receive all baseline measures and questionnaires. Post injection they will receive the primary outcome measures: 1) Numeric Pain Rating Scale and 2) Anxiety thermometer
- Audiovisual (AV) Guided Relaxation (Active Comparator): Combination Product: Audiovisual Guided Relaxation Five-minute guided relaxation delivered via a computer screen and speakers
  Interventions: Combination Product: Audiovisual Guided Relaxation
- Virtual Reality (VR) Guided Relaxation (Experimental): Combination Product: Virtual Reality Guided Relaxation Five-minute guided relaxation delivered via a Samsung Galaxy 7s and the Samsung adaptable VR headset.
  Other Names:
  • Samsung Galaxy 7s/Samsung adaptable VR headset
  Interventions: Combination Product: Virtual Reality Guided Relaxation

INTERVENTIONS:
Combination Product: Audiovisual Guided Relaxation — Five-minute guided relaxation delivered via a computer screen and speakers
  Arms: Audiovisual (AV) Guided Relaxation
Combination Product: Virtual Reality Guided Relaxation — Five-minute guided relaxation delivered via a Samsung Galaxy 7s and the Samsung adaptable VR headset.
  Arms: Virtual Reality (VR) Guided Relaxation

SUMMARY:
The management of chronic pain is a significant public health issue related to escalating treatment costs, lost productivity, disability and medication use. The prevalence of chronic pain is rising alarmingly across all subpopulations with chronic low back pain (LBP) being labeled as one of the 15 most expensive medical conditions. Both study investigators are involved in the medical treatment of these patients. The investigators are interested in testing the effectiveness of alternative treatment strategies that address the complexity of chronic pain that is often mediated not only by physiologic variables, but also psychosocial issues. There is emerging evidence that Virtual Reality (VR) may be an effective pain management tool to augment care in this population, reducing medical costs, decreasing medication use, improving outcomes and empowering patients to take more control over their own health and management of chronic pain. Less is known about the use of this technology delivered in the context of care delivered in an outpatient clinical setting.

DETAILED DESCRIPTION:
The investigators propose to conduct a comparative randomized trial of 45 patients who will be recruited during their office visit at the Spaulding Rehabilitation Hospital Outpatient Center in Cambridge and/or the Massachusetts General Hospital (MGH) Spine Center in Boston. All patients with chronic LBP who elect to receive a spinal injection will be eligible to be screened for inclusion and exclusion criteria. Prior to the injection appointment in Charlestown, Massachusetts, chronic lumbar pain patients are seen by the interventional physiatrist for an examination and discussion of pain management care options. If the patient and MD determine that a spinal injection is indicated, and the patient meets the inclusion criteria, the medical assistant will hand the patient an informational flyer describing study procedures and briefly describe the study. As the study poses minimal risks and low patient time burden beyond the context of standard clinical care, the patient will indicate their wiliness to participate at the end of this clinic visit.

The patient's status will be registered in Epic and will be viewable by authorized study staff. If a consented study participant is active on gateway, the Epic Patient Reported Outcome Information System (PROMIS) measures identified could be administered via the Epic patient portal or they could be administered via iPad as per usual procedures at the injection clinic appointment in Charlestown. Upon arrival to the injection appointment in Charlestown, front desk personnel will hand study participants (flagged in the Epic record) additional paper questionnaires that are not included in the Patient Reported Outcome Measures (PROMs) PROMIS questionnaire battery but are recommended by the National Institute of Health (NIH) task force on research on chronic LBP patients or otherwise identified by the co-investigators as important to address the study aims. If the patient is not active on gateway, an iPad will be used to collect the PROMs PROMIS Epic measures upon clinic arrival. Once all measures have been collected, patients will be randomized using a computer-generated schedule that will randomly assign participants into either the control, computer delivered audiovisual intervention (AV), or the virtual reality (VR) delivered intervention.

Those patients randomized into the control group will receive usual care. After the injection, the control group will receive the anxiety measure and the pain intensity measure. These will be administered in paper format and collected by authorized study personnel. This will conclude study participation.

Study participants randomized into the audiovisual (AV) intervention group will watch and listen to a 5-minute guided relaxation session on a computer in the pre-procedure examination room prior to the injection. The injection is not part of the study procedures and is performed in a separate fluoroscopy suite. Authorized study personnel will be present in the clinic on injection days. Clinic personnel will notify study staff of the patient's randomized status. Study staff will enter the injection preparation room and make sure the patient is comfortably seated. Study staff will launch the 5-minute audiovisual presentation on a computer and leave the room. Clinic personnel will enter after the presentation is concluded and continue with standard clinic preparation for the injection. The presentation is commercially available by Provata Health. No data will be collected or identifying information provided in this process. After receiving the injection and returning to the preparation exam room, study staff will facilitate completion of the anxiety thermometer, the pain intensity measures, and a single response measure that asks if they would be interested in viewing the same presentation on their home computers. This will conclude study participation.

Those study participants randomized into the VR group will watch and listen to the same 5-minute presentation via a VR headset and smart phone. Once a study participant's status has been randomized into the VR group, study staff will enter the injection preparation room, ensure the participant is comfortably seated, orient the participant to the device, apply the headset on the participant to ensure comfort and launch the VR 5-minute presentation. Study staff will then exit the room. No data will be collected or identifying information provided during this process. The Samsung Galaxy 7s and the Samsung adaptable VR headset will be used to deliver the intervention. Clinic staff will enter the room after the 5-minute VR presentation and continue with standard clinic pre-injection procedures. After the injection and upon return to the preparation room, study staff will facilitate administration of the anxiety thermometer measure, the pain intensity measure, the virtual reality symptom questionnaire that addresses 13 symptoms that people who view VR delivered content may experience, and a single response question that asks if they would be interested in viewing the VR content on their own at home. This will conclude study participation.

The VR headset will utilize a disposable cloth face barrier and will be thoroughly cleaned with alcohol solution between patient use. A disposable hygienic face barrier will be applied to all areas of possible direct patient contact of the VR headset. This barrier is held in place by cloth straps, is hypoallergenic, and only surrounds the eyes (therefore will not affect vision or respiration). Provata health produces content that can be delivered through VR or regular delivery via a computer screen (AV). By delivering identical content in two different ways, the investigators will be able to determine if the method of delivery provides any specific advantages or disadvantages. The investigators will also be able to compare outcomes with those who received usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients attending an appointment to receive a lumbar spinal injection.
2. Patients meeting the definition of chronic LBP as established by the NIH task force: Back pain problem that has persisted at least 3 months, and has resulted in pain on at least half the days in the past 6 months

Exclusion Criteria:

1. Age younger than 18 years
2. Not being fluent and literate in English
3. Patients receiving injections in areas other than the lumbar or pelvic region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change is being assessed between two time points by The Numeric Pain Rating Scale | First time point: At the beginning of the injection clinic visit, prior to receiving the injection. Second time point: approximately 1 hour later, at the conclusion of the injection clinic visit, after receiving the injection
  Self-report current pain rating on a 0-10 scale with 0 being no pain and 10 being the worst pain imaginable

SECONDARY OUTCOMES:
Change is being assessed between two time points by The Anxiety Thermometer | First time point: At the beginning of the injection clinic visit, prior to receiving the injection. Second time point: approximately 1 hour later, at the conclusion of the injection clinic visit, after receiving the injection
  a visual numeric rating scale of current anxiety level from 0-10 with 0 being not at all anxious up to 10 being extremely anxious
Virtual Reality Symptom Questionnaire | Measured at one time point approximately 1 hour from the time of randomization
  This is a self report measure related to symptoms encountered when viewing virtual reality content. This questionnaire will only be administered to the participants randomized into the virtual reality group. Description: 13 symptoms are rated from 0-6 with 0 being no symptoms; 1-2=slight; 3-4=moderate; 5-6=severe; the 13 categories are: general discomfort, fatigue, boredom, drowsiness, headache, dizziness, difficulty concentrating, nausea, sore/aching eyes, tired eyes, eye strain, blurred vision, difficulty focusing; scored as a sum of all categories

OTHER OUTCOMES:
Interest questions about the guided relaxation content | Measured at one time point approximately 1 hour from the time of randomization
  This questionnaire will be administered to those participants randomized into the audiovisual and the virtual reality groups. 1. Would you be interested in having the guided relaxation video to view:
  i. On your computer at home? ii. On a VR headset at home? 2. Do you feel this type of guided relaxation might be useful in helping you manage your pain?

CONTACTS AND LOCATIONS:
Overall Officials: David S Binder, MD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ames SL, Wolffsohn JS, McBrien NA. The development of a symptom questionnaire for assessing virtual reality viewing using a head-mounted display. Optom Vis Sci. 2005 Mar;82(3):168-76. doi: 10.1097/01.opx.0000156307.95086.6. PMID 15767873
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Background] Chan E, Foster S, Sambell R, Leong P. Clinical efficacy of virtual reality for acute procedural pain management: A systematic review and meta-analysis. PLoS One. 2018 Jul 27;13(7):e0200987. doi: 10.1371/journal.pone.0200987. eCollection 2018. PMID 30052655
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Dascal J, Reid M, IsHak WW, Spiegel B, Recacho J, Rosen B, Danovitch I. Virtual Reality and Medical Inpatients: A Systematic Review of Randomized, Controlled Trials. Innov Clin Neurosci. 2017 Feb 1;14(1-2):14-21. eCollection 2017 Jan-Feb. PMID 28386517
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Houtman IL, Bakker FC. The anxiety thermometer: a validation study. J Pers Assess. 1989 Fall;53(3):575-82. doi: 10.1207/s15327752jpa5303_14. PMID 2778618
- [Background] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. 2015 Feb 18;350:h444. doi: 10.1136/bmj.h444. PMID 25694111
- [Background] Westenberg RF, Zale EL, Heinhuis TJ, Ozkan S, Nazzal A, Lee SG, Chen NC, Vranceanu AM. Does a Brief Mindfulness Exercise Improve Outcomes in Upper Extremity Patients? A Randomized Controlled Trial. Clin Orthop Relat Res. 2018 Apr;476(4):790-798. doi: 10.1007/s11999.0000000000000086. PMID 29480886
- See also: Institute of Medicine (US) Committee on Advancing Pain Research,Care, and Education. (2011). Relieving {Pain} in {America}: {A} {Blueprint} for{Transforming} {Prevention}, {Care}, {Education}, and {Research}. — http://www.ncbi.nlm.nih.gov/books/NBK91497/
- See also: Kamper, S. J., Apeldoorn, A. T., Chiarotto, A., Smeets, R. J. E. M.,Ostelo, R. W. J. G., Guzman, J., & Tulder, M. W. V. (2015). Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ — http://doi.org/10.1136/bmj.h444